CLINICAL TRIAL: NCT04340960
Title: Effect of Continuity of Care With Digital Home Monitoring on Postoperative Outcomes in Patients Undergoing Thoracic Surgery: A Pilot Randomized Controlled Trial (CDHM: RCT)
Brief Title: Home Monitoring for Thoracic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Yamini Subramani, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDHM:RCT
Record Dates: First submitted 2020-03-24; First posted 2020-04-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will not be monitored with continuity of care. After this period, 30-day emergency department visits will be measured and compared between the two groups, along with 30-day readmission rates, in-hospital length of stay, mortality, quality of recovery 40 item scale (QoR-40), European Quality of Life 5 Dimensions (EQ5D), patient satisfaction score, and societal and hospital cost.
  No intervention will be administered.
- Home Monitoring Group (Experimental): At the time of hospital discharge, the control group will be discharged without receipt of home monitoring, and the intervention group will receive a home monitoring kit with (NIBP (non-invasive blood pressure) and SPO2 (pulse oximetry) with instructions on how to use these devices. Patients in the intervention groups will receive digital communication for four weeks and have their NIBP, HR (heart rate), SPO2 and pain scores evaluated twice a day for two weeks.
  Interventions: Other: Home Monitoring

INTERVENTIONS:
Other: Home Monitoring — Patients in this group will receive home monitoring for NIBP (non-invasive blood pressure), SPO2 (pulse oximetry), and pain scores. These will be monitored 4 times a day for 2 weeks following surgery.
  Arms: Home Monitoring Group

SUMMARY:
Background and Importance: When patients transition from hospital to home following surgery, perceived complications or poorly controlled pain can result in emergency department visits and readmissions. Continuity of care after discharge has been shown to reduce ED visits and readmissions rates. Hence any improved method of extending the continuity of care in a patient's home may improve postoperative outcomes. For patients who are at risk, continuity of care with digital solutions offers a pathway to providing more education, influencing behaviour, and creating better outcomes. Care teams can understand what's going on with each patient daily or weekly, as opposed to sporadically through an office visit.

Goals/Research Aims: Atrial fibrillation is one of the important complications after thoracic surgery, it is estimated to occur in 10.5% of patients. We will conduct a randomized controlled trial to test the use of a secured digital system to monitor vital signs and home-based ECG monitoring for 2 weeks after surgery in patients undergoing an elective thoracic surgical procedure at the London Health Sciences Centre [LHSC]. Specific objectives are to determine the feasibility of 30-day emergency department visits as the primary outcome, 30-day readmission rates, postoperative complications, in-hospital length of stay, pain scores, hospital case costing, societal costs, mortality, and patient satisfaction.

Methods/Approaches/Expertise: This trial will be a single centre, assessor-blinded, parallel arm, randomized controlled trial. Participants will be recruited from patients scheduled for thoracic surgical procedures at LHSC. Patients will be randomized to either the Continuity of care with Digital Home Monitoring (CDHM) group or the control group. The control group will be provided with the usual post-operative care, and the CDHM group will be provided with access to self-help resources, digital monitoring and access to a clinical navigator for two weeks. All outcomes will be compared between the CDHM group and control group at the end of 4 weeks post-discharge, including out-of-pocket costs, travel costs and lost productivity.

Expected Outcomes: The Ontario Hospital Association estimates the average cost of a one-day stay in an acute care hospital is $1,300. With digital monitoring and continuity of care, we expect to decrease visits and readmission rates by at least 50% and in-hospital length stay by at least one day. This is a feasibility study. We will follow the traffic light approach criteria for reporting feasibility outcomes: Feasible (green) 75-100%: all feasibility outcomes are met; no protocol modifications are needed; (2) Feasible with modification (amber) 50-75%: all feasibility outcomes are met or can be met with protocol modifications; (3) Not feasible (red) <50%: even with protocol modifications, some feasibility outcome cannot be met.

DETAILED DESCRIPTION:
Introduction: Surgical recovery after discharge from the hospital often poses confusion and challenges for patients and caregivers. This is more so when early dismissal after surgery has become the norm. Furthermore, the Canadian health care system is fragmented, with poorly integrated services. Thus, when patients transition from hospital to home following surgery, complications and inadequately controlled pain results in return to hospital or ED visits. Family caregivers are frustrated that health care providers involved in different aspects of a patient's care do not always communicate with one another, resulting in caregivers having to retell a patient's story and spending unnecessary time clarifying information during the ED visits. Caregivers and healthcare providers are looking for one clear point of contact that ensures patients' needs are met at every segment of their healthcare journey. Patients believe that when they receive care, it is generally of high quality. Despite the positive feedback from the patients about the quality of care, the system continues to struggle with transitional care due to a lack of system-wide integration.

This randomized controlled trial on continuity of care with digital home monitoring for four weeks post-operatively in patients undergoing an elective thoracic surgical procedure.

Eligible patients will be recruited from the surgeon's office, and informed consent will be obtained. Patients will be randomized to the control group (no digital care) or the intervention groups (digital care provided). Intraoperative and immediate postoperative care in the post-anesthesia care unit (PACU) and surgical ward will remain the same for all patients. At the time of hospital discharge, the control group will be discharged without receipt of home monitoring, and the intervention group will receive a home monitoring kit with (NIBP (non-invasive blood pressure) and SPO2 (pulse oximetry) with instructions on how to use these devices. Patients in the intervention groups will receive digital communication for four weeks and have their NIBP, HR (heart rate), SPO2 and pain scores evaluated once a day for two weeks. The control group will not be monitored with continuity of care. After this period, 30-day emergency department visits will be measured and compared between the two groups, along with 30-day readmission rates, in-hospital length of stay, mortality, quality of recovery 40 item scale (QoR-40), European Quality of Life 5 Dimensions (EQ5D), patient satisfaction score, and societal and hospital cost.

ED visits and readmission rate: In Ontario, between 2014 and 2016, within 30 days after lung cancer lobectomy surgery, the readmission rate was 5.9%, and the Emergency Department (ED) visit rate was 16.2%.(1) At the LHSC, the 30-day ED visit rates were 21.5% [95% CI 15.91, 27.14], and the 30-day readmission rates were 6.73% [95% CI 3.21, 10.24] for lung cancer lobectomy.(1) Between 2015/2016 and 2017/2018, unadjusted data of readmissions or ED visits within seven days after Video Assisted Thoracoscopic Surgery (VATS) and open thoracotomy were 9% and 7%, respectively, at LHSC. Post-surgical discharge hospital visits remain a significant problem in post-thoracic surgical care. Patients have to wait too long during ED visits, which negatively impacts provider, caregiver and patient well-being. The investigators believe that a virtual care option extending the continuity of care post-discharge is a viable solution to this problem.

Digital solution - virtual care: In the last few years, the focus on patient care has moved from clinical to home. Now, more than ever, it is necessary to engage patients before, throughout the perioperative period, and in rehabilitation, post-surgery to ensure the best possible patient health outcomes while reducing LOS and unplanned readmissions. Ensuring patients are prepared to adhere to the post-surgical plan of care once released from the hospital can increase the length of hospital stay by as much as 25%. Digital solutions can alleviate the problem by enabling remote monitoring of a patient's vital signs, symptoms and behaviour at home, sending medication reminders, monitoring medication use and the patient's understanding of the self-care content it is delivering, ensuring patients remain on the pathway toward better health, finally improving the patient's outcomes.

Continuity of care: Continuity of care after discharge has been shown to reduce readmissions and ED visits. Hence, extending the continuity of care in a patient's home may reduce revisit rates. (2) In one study on thoracic surgery, 30-day readmissions were reduced using a hospital-operated "Integrated Comprehensive Care" program, comprised of a single nurse coordinator, eight registered and practical nurses, and six physiotherapists, along with respiratory therapists, dieticians, and occupational therapists on an "as-needed" basis. (3) In another study, education, coordinated discharge, physician follow-up, & home visits all contributed to reduced readmission rates. (4) Of note, Canadian data show that within the first seven days after surgical discharge, 28.3% of the diagnoses fall within the Canadian Emergency Department Triage and Acuity Scale (CTAS) IV or V; i.e. less or non-urgent. Those are likely manageable at the patient's home if appropriate transitional care is available and possibly preventable.

For patients at risk or rising at risk, continuity of care with digital solutions offers a pathway to providing more education, influencing behaviour, and creating better outcomes for patient populations. Care teams can understand what's going on with each patient daily or weekly, as opposed to once or twice a year through an office visit. With a continuous and more complete picture of patient health, they can adjust care plans as needed and proactively engage populations in managing their care.

ECG monitoring: The investigators incorporated home-based ECG monitoring in this population because atrial fibrillation is one of the critical indicators of adverse outcomes after thoracic surgery. After thoracic surgery, postoperative atrial fibrillation (POAF) occurs in 10.5% of patients(4), 7.3% after Video-Assisted Thoracoscopic Surgery (VATS) and 11.7% in open thoracotomy. (5) In major non-cardiac surgery as a group, the incidence of POAF is 3.0% (6), making POAF, after thoracic surgery, one of the highest in non-cardiac surgery. POAF is associated with infections (7); increased mortality (6); intra-operative transfusions (8); post-operative transfusions (9); post-operative pneumonia (10); respiratory failure (11); and therefore may be an important sign, or result, of postoperative complications, rather than the cause. In one study, POAF occurred at a mean of 3.55 days, with an increased in-hospital length of stay [LOS]. (7) Long-term follow-up of over 900 days showed that POAF recurs in 17.1% of non-cardiac surgical patients, with implications for long-term cerebrovascular accidents (CVA). (12) In a database study of 1,729,360 patients, POAF in non-cardiac surgery was associated with a CVA within one year, at an HR of 2.0 (1.7 - 2.3) compared to cardiac surgery or a cumulative rate of 1.47% (95% CI 1.24 - 1.75%). (13) Associated with higher mortality and complications, POAF adds another dimension to the high rate of unplanned hospital visits after thoracic surgical discharge.

Digital Monitoring: Even though continuous monitoring is the standard of care in the postanesthesia care unit, patients are managed by periodic vital checks by the nursing team in the surgical wards and no monitoring after the hospital discharge. Once patients are discharged from the hospital, patients and family caregivers feel vulnerable and abandoned. Digital home monitoring and digital self-care, such as blood pressure and SPO2 measurement at home, enable a small number of providers to coach many patients. Post-operative home monitoring with non-invasive blood pressure (NIBP), heart rate (HR), hemoglobin oxygen saturation (SpO2), & pain scores collected at regular intervals has been instituted previously. (14) Such monitoring will help stratify CTAS IV/V patients from CTAS I, II, or III cases. Along with the vitals, home-based ECG monitoring will allow detection of early signs and symptoms of any concerns, which can be intervened and managed remotely.

The proposed trial:

Therefore, the investigators propose a pilot randomized controlled trial on continuity of care with digital home monitoring for two weeks post-operatively in patients undergoing an elective thoracic surgical procedure and four weeks of two-way communication.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to provide informed consent
* Availability of a caregiver at the patient's home
* Wi-fi or cellular connectivity at the patient's home
* Undergoing elective segmentectomy, lobectomy, or pneumonectomy; VATS or open procedure and any thoracic foregut procedure like esophagectomy etc
* ASA III or lower
* Ability to comprehend and consent in English
* Patient or caregiver familiar/comfortable with the use of the technology like online banking

Exclusion Criteria:

* Unstable disease process preoperatively
* Patient requiring postoperative ICU admission
* Expected unstable disease process in the postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Trial Recruitment | 1 year
  Number of patients recruited over the period of the study, a measure of study feasibility
Protocol adherence | 1 year
  As collected on the Case Report Forms and loss-to-follow-up
Outcome data collection | 1 year
  Data will be collected from the patient on the vitals and daily assessment on the video call.

SECONDARY OUTCOMES:
Patient satisfaction score | 30 days postoperatively
  Using 5 point Likert's satisfaction scale: a 5-point Likert scale, 1 - strongly disagree, 2 - disagree, 3 - neutral, 4 - agree and 5 - strongly agree,
Patient/caregiver experience | 30 days postoperatively
  Using 5 point Likert's satisfaction scale: a 5-point Likert scale, 1 - strongly disagree, 2 - disagree, 3 - neutral, 4 - agree and 5 - strongly agree,
30 day ED visit; 30 day readmission rate; cost analysis etc | 30 days postoperatively
  Thirty day hospital readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Yamini Subramani, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Book. All-Cause Readmission to Acute Care and Return to the Emergency Department. Ottawa, ON. Canadian Institute for Health Information. 2012 ISBN: 978-1-77109-040-7. :Available from: https://secure.cihi.ca/free_produc.
- [Background] MOH. June 2019 report of the Premier's Council on Improving Healthcare and Ending Hallway Medicine: "Healthy Ontario: Building a Sustainable Health Care System.
- [Background] Yang H, Dervin G, Madden S, Beaulé P, Gagné S, Crossan M, Fayad A, Wheeler K, Afagh M, Zhang T, Taljaard M. Post-Op Home Monitoring after Joint Replacement (POHM): A feasibility study. Innov Fund Prov Overs Comm Showc 2016; Toronto, ON Canada2016.
- [Background] Cancer Care Council of Ontario. Unplanned Hospital Visits After Surgery. :Available from: http://www.csqi.on.ca/by_patient_j.
- [Background] van Walraven C, Mamdani M, Fang J, Austin PC. Continuity of care and patient outcomes after hospital discharge. J Gen Intern Med. 2004 Jun;19(6):624-31. doi: 10.1111/j.1525-1497.2004.30082.x. PMID 15209600
- [Background] Shargall Y, Hanna WC, Schneider L, Schieman C, Finley CJ, Tran A, Demay S, Gosse C, Bowen JM, Blackhouse G, Smith K. The Integrated Comprehensive Care Program: A Novel Home Care Initiative After Major Thoracic Surgery. Semin Thorac Cardiovasc Surg. 2016 Summer;28(2):574-582. doi: 10.1053/j.semtcvs.2015.12.003. Epub 2015 Dec 11. PMID 28043480
- [Background] Young JM, Butow PN, Walsh J, Durcinoska I, Dobbins TA, Rodwell L, Harrison JD, White K, Gilmore A, Hodge B, Hicks H, Smith S, O'Connor G, Byrne CM, Meagher AP, Jancewicz S, Sutherland A, Ctercteko G, Pathma-Nathan N, Curtin A, Townend D, Abraham NS, Longfield G, Rangiah D, Young CJ, Eyers A, Lee P, Fisher D, Solomon MJ. Multicenter randomized trial of centralized nurse-led telephone-based care coordination to improve outcomes after surgical resection for colorectal cancer: the CONNECT intervention. J Clin Oncol. 2013 Oct 1;31(28):3585-91. doi: 10.1200/JCO.2012.48.1036. Epub 2013 Sep 3. PMID 24002519
- [Background] Jeon JH, Kang CH, Kim HS, Seong YW, Park IK, Kim YT, Kim JH. Video-assisted thoracoscopic lobectomy in non-small-cell lung cancer patients with chronic obstructive pulmonary disease is associated with lower pulmonary complications than open lobectomy: a propensity score-matched analysis. Eur J Cardiothorac Surg. 2014 Apr;45(4):640-5. doi: 10.1093/ejcts/ezt460. Epub 2013 Sep 19. PMID 24052605
- [Background] Cao C, Zhu ZH, Yan TD, Wang Q, Jiang G, Liu L, Liu D, Wang Z, Shao W, Black D, Zhao Q, He J. Video-assisted thoracic surgery versus open thoracotomy for non-small-cell lung cancer: a propensity score analysis based on a multi-institutional registry. Eur J Cardiothorac Surg. 2013 Nov;44(5):849-54. doi: 10.1093/ejcts/ezt406. Epub 2013 Aug 15. PMID 23956268
- [Background] Bhave PD, Goldman LE, Vittinghoff E, Maselli J, Auerbach A. Incidence, predictors, and outcomes associated with postoperative atrial fibrillation after major noncardiac surgery. Am Heart J. 2012 Dec;164(6):918-24. doi: 10.1016/j.ahj.2012.09.004. Epub 2012 Oct 26. PMID 23194493
- [Background] Garner M, Routledge T, King JE, Pilling JE, Veres L, Harrison-Phipps K, Bille A, Harling L. New-onset atrial fibrillation after anatomic lung resection: predictive factors, treatment and follow-up in a UK thoracic centre. Interact Cardiovasc Thorac Surg. 2017 Feb 1;24(2):260-264. doi: 10.1093/icvts/ivw348. PMID 27803121
- [Background] Vaporciyan AA, Correa AM, Rice DC, Roth JA, Smythe WR, Swisher SG, Walsh GL, Putnam JB Jr. Risk factors associated with atrial fibrillation after noncardiac thoracic surgery: analysis of 2588 patients. J Thorac Cardiovasc Surg. 2004 Mar;127(3):779-86. doi: 10.1016/j.jtcvs.2003.07.011. PMID 15001907
- [Background] Imperatori A, Mariscalco G, Riganti G, Rotolo N, Conti V, Dominioni L. Atrial fibrillation after pulmonary lobectomy for lung cancer affects long-term survival in a prospective single-center study. J Cardiothorac Surg. 2012 Jan 10;7:4. doi: 10.1186/1749-8090-7-4. PMID 22233837
- [Background] Amar D, Zhang H, Leung DH, Roistacher N, Kadish AH. Older age is the strongest predictor of postoperative atrial fibrillation. Anesthesiology. 2002 Feb;96(2):352-6. doi: 10.1097/00000542-200202000-00021. PMID 11818768
- [Background] Ayoub K, Habash F, Almomani A, Xu J, Marji M, Shaw-Devine A, Paydak H, Vallurupalli S. Long Term Risk of Recurrent Atrial Fibrillation and Ischemic Stroke after Post-Operative Atrial Fibrillation Complicating Cardiac and Non-Cardiac Surgeries. J Atr Fibrillation. 2018 Apr 30;10(6):1660. doi: 10.4022/jafib.1660. eCollection 2018 Apr. PMID 29988296
- [Background] Gialdini G, Nearing K, Bhave PD, Bonuccelli U, Iadecola C, Healey JS, Kamel H. Perioperative atrial fibrillation and the long-term risk of ischemic stroke. JAMA. 2014 Aug 13;312(6):616-22. doi: 10.1001/jama.2014.9143. PMID 25117130
- [Background] Yang H, Dervin G, Madden S, Beaule PE, Gagne S, Crossan ML, Fayad A, Wheeler K, Afagh M, Zhang T, Taljaard M. Postoperative Home Monitoring After Joint Replacement: Feasibility Study. JMIR Perioper Med. 2018 Sep 5;1(2):e10168. doi: 10.2196/10168. PMID 33401364
- [Derived] Nagappa M, Subramani Y, Yang H, Wood N, Querney J, Fochesato LA, Nguyen D, Fatima N, Martin J, John-Baptiste A, Nayak R, Qiabi M, Inculet R, Fortin D, Malthaner R. Enhancing Quadruple Health Outcomes After Thoracic Surgery: Feasibility Pilot Randomized Controlled Trial Using Digital Home Monitoring. JMIR Perioper Med. 2025 Feb 12;8:e58998. doi: 10.2196/58998. PMID 39938882